CLINICAL TRIAL: NCT00433537
Title: A Phase II Study of VcR-CVAD With Rituximab Maintenance for Untreated Mantle Cell Lymphoma
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02966; NCI-2012-02966 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E1405 (Other: Eastern Cooperative Oncology Group (ECOG)); E1405 (Other: Eastern Cooperative Oncology Group); E1405 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-01

CONDITIONS: Contiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Stage I Mantle Cell Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Dexamethasone; Calcium Dobesilate; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VcR-CVAD induction followed by maintenance rituximab (Experimental): VcR-CVAD induction: Patients receive VcR-CVAD comprising bortezomib IV over 3-5 seconds on days 1 and 4; rituximab IV over 3-4 hours on day 1; doxorubicin hydrochloride IV over 48 hours on days 1 and 2; cyclophosphamide IV over 3 hours every 12 hours on days 1-3; vincristine IV over 3-5 seconds on day 3; and dexamethasone IV or orally once daily on days 1-4. Patients also receive filgrastim (G-CSF) subcutaneously (SC) or IV once daily beginning on day 5 or 6 and continuing until blood counts recover OR pegfilgrastim SC on day 5 or 6. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance rituximab: Beginning 4-8 weeks after completion of induction therapy, patients receive rituximab IV over 3-4 hours once weekly for 4 weeks. Treatment repeats every 6 months for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine; Drug: dexamethasone; Biological: filgrastim; Biological: pegfilgrastim
- VcR-CVAD induction followed by ASCT (Experimental): VcR-CVAD induction: Patients receive VcR-CVAD comprising bortezomib IV over 3-5 seconds on days 1 and 4; rituximab IV over 3-4 hours on day 1; doxorubicin hydrochloride IV over 48 hours on days 1 and 2; cyclophosphamide IV over 3 hours every 12 hours on days 1-3; vincristine IV over 3-5 seconds on day 3; and dexamethasone IV or orally once daily on days 1-4. Patients also receive filgrastim (G-CSF) SC or IV once daily beginning on day 5 or 6 and continuing until blood counts recover OR pegfilgrastim SC on day 5 or 6. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  ASCT: After completion of induction therapy, patients who are eligible may have the option to receive consolidation therapy for autologous stem cell transplantation (off-study). These patients undergo stem cell harvest during courses 4, 5, or 6 of induction therapy.
  Interventions: Drug: bortezomib; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine; Drug: dexamethasone; Biological: filgrastim; Biological: pegfilgrastim; Procedure: Autologous stem cell transplantation (ASCT)

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine — Given IV
  Other Names: Vincristine sulfate; Leurocristine sulfate; VCR; Vincasar PFS
Drug: dexamethasone — Given IV
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
Procedure: Autologous stem cell transplantation (ASCT)
  Arms: VcR-CVAD induction followed by ASCT

SUMMARY:
This phase II trial is studying how well giving rituximab together with combination chemotherapy and bortezomib works in treating patients with untreated mantle cell lymphoma. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving rituximab together with combination chemotherapy and bortezomib may kill more cancer cells.

Treatment consists of six agents: bortezomib (Vc), rituximab (R), cyclophosphamide (C), vincristine (V), doxorubicin (A), and dexamethasone (D) (VcR-CVAD).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete response (CR) rate in patients with mantle cell lymphoma, who are treated with VcR-CVAD.

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate to VcR-CVAD. II. To evaluate the progression-free survival (PFS) and overall survival (OS) of patients receiving maintenance rituximab after VcR-CVAD induction.

III. To evaluate the PFS and OS of patients who receive autologous stem cell transplantation (ASCT) after VcR-CVAD induction.

IV. To evaluate the toxicity of VcR-CVAD.

TERTIARY OBJECTIVES:

I. Evaluation of antigen expression patterns to determine or confirm possible unique expressions of MCL.

II. To evaluate the percentage of circulating mantle cell lymphoma (MCL) cells.

OUTLINE: This is a multicenter study.

Induction therapy (VcR-CVAD): Patients receive VcR-CVAD comprising bortezomib 1.3 mg/m2 IV over 3-5 seconds on days 1 and 4; rituximab 375 mg/m2 IV over 3-4 hours on day 1; doxorubicin hydrochloride 25 mg/m2/d IV over 48 hours on days 1 and 2; cyclophosphamide 300 mg/m2 IV over 3 hours every 12 hours on days 1-3; vincristine 1 mg IV over 3-5 seconds on day 3; and dexamethasone 40 mg IV or orally once daily on days 1-4. Patients also receive filgrastim (G-CSF) subcutaneously (SC) or IV once daily beginning on day 5 or 6 and continuing until blood counts recover OR pegfilgrastim SC on day 5 or 6. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Maintenance therapy: Beginning 4-8 weeks after completion of induction therapy, patients receive rituximab IV over 3-4 hours once weekly for 4 weeks. Treatment repeats every 6 months for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of induction therapy, patients who are eligible may have the option to receive consolidation therapy for autologous stem cell transplantation (ASCT) (off-study). These patients undergo stem cell harvest during courses 4, 5, or 6 of induction therapy.

After completion of study treatment, patients are followed periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of mantle cell lymphoma by demonstrating appropriate morphology plus at least one of the following on the biopsy specimen: nuclear cyclin D1+ by immunohistochemistry; t(11;14) by fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR), or conventional karyotyping
* No prior chemotherapy, immunotherapy or radiotherapy for mantle cell lymphoma; a brief course of steroids (< 14 days) for symptom relief or steroids for other indications are allowed
* Patients must have measurable disease; CT scans at baseline are required to define the extent of measurable disease; the scans must be obtained within 6 weeks prior to registration; combined CT/PET scans may be used for the baseline and subsequent evaluations if accurate tumor measurements can be obtained from the CT component
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) > 1500 mm^3 (unless low count due to marrow involvement or splenomegaly)
* Platelets > 100,000 mm^3 (unless low counts due to marrow involvement or splenomegaly)
* Creatinine < 2 mg/dL
* Bilirubin < 2 mg/dL (may be up to 3.0 mg/dL if due to Gilbert's disease or due to liver involvement by lymphoma)
* Patients over the age of 45 must have a left ventricular ejection fraction (LVEF) of greater than 45% documented within 90 days prior to registration
* Patients must be tested for Hepatitis B surface antigen (HBs Ag) within 4 weeks prior to registration NOTE: HBs Ag positive patients are not excluded but will have more stringent monitoring of liver function tests

Exclusion Criteria:

* Known HIV disease; an HIV test is not required for entry on study but is required if the patient is perceived to be at risk; patients with a history of intravenous drug use or any other behavior with an increased risk for HIV infection should be tested for exposure to the HIV virus; patients with known HIV are excluded since the immunocompromised state of patients with HIV infection or the concomitant use of highly active antiretroviral therapy (HAART) may result in more extensive dose modifications than intended for the intensive therapeutic regimen used in this study
* Pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; women of childbearing potential and sexually active males must use an accepted and effective method of contraception
* Grade 2 or higher baseline peripheral neuropathy
* Known hypersensitivity to boron or mannitol
* History of prior malignancy unless at least one of the following conditions are met:

  * Malignancy was in-situ
  * Malignancy was treated surgically or with local radiation therapy with curative intent and the patient has been disease free for > 3 years
  * Any adjuvant hormonal therapy must have been discontinued > 3 months prior to registration
* Known central nervous system (CNS) involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kahl, Study Chair — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chang JE, Li H, Smith MR, Gascoyne RD, Paietta EM, Yang DT, Advani RH, Horning SJ, Kahl BS. Phase 2 study of VcR-CVAD with maintenance rituximab for untreated mantle cell lymphoma: an Eastern Cooperative Oncology Group study (E1405). Blood. 2014 Mar 13;123(11):1665-73. doi: 10.1182/blood-2013-08-523845. Epub 2014 Jan 23. PMID 24458437

RESULTS

PARTICIPANT FLOW:
Groups:
- VcR-CVAD Induction Followed by Maintenance Rituximab: VcR-CVAD induction: Patients receive VcR-CVAD comprising bortezomib IV over 3-5 seconds on days 1 and 4; rituximab IV over 3-4 hours on day 1; doxorubicin hydrochloride IV over 48 hours on days 1 and 2; cyclophosphamide IV over 3 hours every 12 hours on days 1-3; vincristine IV over 3-5 seconds on day 3; and dexamethasone IV or orally once daily on days 1-4. Patients also receive filgrastim (G-CSF) subcutaneous (SC) or IV once daily beginning on day 5 or 6 and continuing until blood counts recover OR pegfilgrastim SC on day 5 or 6. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance rituximab: Beginning 4-8 weeks after completion of induction therapy, patients receive rituximab IV over 3-4 hours once weekly for 4 weeks. Treatment repeats every 6 months for up to 4 courses in the absence of disease progression or unacceptable toxicity.
- VcR-CVAD Induction Then Off Study: Patients received VcR-CVAD induction but did not proceed to step 2 treatment for various reasons.
Period: Step 1 - VcR-CVAD Induction
Arm/Group | VcR-CVAD Induction Followed by Maintenance Rituximab | VcR-CVAD Induction Followed by ASCT | VcR-CVAD Induction Then Off Study
Started | 45 | 22 | 10
Eligible and Treated | 44 | 22 | 9
Completed | 44 | 22 | 1
Not Completed | 1 | 0 | 9
Not completed — Path ineligible (not having MCL) | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Period: Step 2 - Maintenance Rituximab or ASCT
Arm/Group | VcR-CVAD Induction Followed by Maintenance Rituximab | VcR-CVAD Induction Followed by ASCT | VcR-CVAD Induction Then Off Study
Started | 45 (This included all treated patients regardless of eligibility.) | 22 | 0 (One patient completed VcR-CVAD and then withdrew from the study.)
Eligible and Treated | 44 | 22 | 0
Completed | 29 | 22 | 0
Not Completed | 16 | 0 | 0
Not completed — Path ineligible (not having MCL) | 1 | 0 | 0
Not completed — Lack of Efficacy | 8 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Alternative therapy | 4 | 0 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients who received VcR-CVAD induction.
Groups:
- Step 1 - VcR-CVAD Induction: All eligible patients who received VcR-CVAD induction.
Arm/Group | Step 1 - VcR-CVAD Induction
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Number of eligible, treated participants who achieve complete response. Response criteria are based upon the criteria from the Revised Response Criteria for Malignant Lymphoma (Cheson et al., 2007). Complete response is defined as complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy.
Time Frame: Assessed after VcR-CVAD cycles 2, 4, and 6.
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion
Groups:
- VcR-CVAD Induction: All eligible patients who received VcR-CVAD induction.
Arm/Group | VcR-CVAD Induction
Number analyzed (Participants) | 75
proportion | 0.68 [0.57 to 0.79]

2. Secondary Outcome: 2-year Progression-free Survival (PFS)
Description: PFS for patients who received maintenance rituximab or ASCT after VcR-CVAD induction is defined as time from start of maintenance rituximab or ASCT to earlier of disease progression or death. Patients alive and progression-free at last follow-up were censored.
Time Frame: Assessed every 6 months for 5 years, and then yearly thereafter.
Population: Eligible and treated patients who received maintenance rituximab or ASCT
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- VcR-CVAD Induction Followed by Maintenance Rituximab: VcR-CVAD induction: Patients receive VcR-CVAD comprising bortezomib IV over 3-5 seconds on days 1 and 4; rituximab IV over 3-4 hours on day 1; doxorubicin hydrochloride IV over 48 hours on days 1 and 2; cyclophosphamide IV over 3 hours every 12 hours on days 1-3; vincristine IV over 3-5 seconds on day 3; and dexamethasone IV or orally once daily on days 1-4. Patients also receive filgrastim (G-CSF) SC or IV once daily beginning on day 5 or 6 and continuing until blood counts recover OR pegfilgrastim SC on day 5 or 6. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance rituximab: Beginning 4-8 weeks after completion of induction therapy, patients receive rituximab IV over 3-4 hours once weekly for 4 weeks. Treatment repeats every 6 months for up to 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | VcR-CVAD Induction Followed by Maintenance Rituximab | VcR-CVAD Induction Followed by ASCT
Number analyzed (Participants) | 44 | 22
probability | 0.79 [0.67 to 0.92] | 0.76 [0.58 to 1]

3. Secondary Outcome: 3-year Overall Survival (OS)
Description: OS for patients who received maintenance rituximab or ASCT after VcR-CVAD induction is defined as time from start of maintenance rituximab or ASCT to death. Patients alive at last follow-up were censored.
Time Frame: Assessed every 6 months for 5 years, and then yearly thereafter.
Population: Eligible and treated patients who received maintenance rituximab or ASCT
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | VcR-CVAD Induction Followed by Maintenance Rituximab | VcR-CVAD Induction Followed by ASCT
Number analyzed (Participants) | 44 | 22
probability | 0.91 [0.83 to 1] | 0.96 [0.87 to 1]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Description: Autologous stem cell transplantation (ASCT) was optional for this study, and submission of data with details on conditioning regimen or toxicity was not mandated. Therefore, the adverse event table for ASCT arm was not available.
Groups:
- Step 1 - VcR-CVAD Induction: All patients who received VcR-CVAD induction.
- Step 2 - Maintenance Rituximab: All patients who received maintenance rituximab.
Arm/Group | Step 1 - VcR-CVAD Induction | Step 2 - Maintenance Rituximab
Serious Adverse Events (participants affected / at risk) | 72/77 | 16/45
Other Adverse Events (participants affected / at risk) | 76/77 | 40/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - VcR-CVAD Induction (N=77) | Step 2 - Maintenance Rituximab (N=45)
Allergic reaction (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 22 | 1
Leukocytes decreased (Investigations) | 52 | 3
Lymphopenia (Investigations) | 50 | 12
Neutrophils decreased (Investigations) | 62 | 7
Platelets decreased (Investigations) | 49 | 0
Hematologic-other (Blood and lymphatic system disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Fatigue (General disorders) | 8 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Weight gain (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 0
Infection w/ gr3-4 neut, catheter relate (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, catheter (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, heart (Infections and infestations) | 0 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 2 | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, blood (Infections and infestations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 1 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Cystitis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - VcR-CVAD Induction (N=77) | Step 2 - Maintenance Rituximab (N=45)
Anemia (Blood and lymphatic system disorders) | 71 | 26
Leukocytes decreased (Investigations) | 39 | 21
Lymphopenia (Investigations) | 39 | 27
Neutrophils decreased (Investigations) | 34 | 12
Platelets decreased (Investigations) | 67 | 19
Hematologic-other (Blood and lymphatic system disorders) | 4 | 0
Hypotension (Vascular disorders) | 5 | 0
Fatigue (General disorders) | 65 | 13
Fever w/o neutropenia (General disorders) | 6 | 0
Insomnia (Psychiatric disorders) | 19 | 0
Rigors/chills (General disorders) | 6 | 0
Weight gain (Investigations) | 6 | 0
Weight loss (Investigations) | 7 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 6
Nail changes (Skin and subcutaneous tissue disorders) | 4 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 | 0
Anorexia (Metabolism and nutrition disorders) | 25 | 0
Constipation (Gastrointestinal disorders) | 41 | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 21 | 0
Dyspepsia (Gastrointestinal disorders) | 10 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 5 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 12 | 0
Nausea (Gastrointestinal disorders) | 53 | 0
Taste disturbance (Nervous system disorders) | 11 | 0
Vomiting (Gastrointestinal disorders) | 23 | 0
Edema limb (General disorders) | 19 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 0
Alkaline phosphatase increased (Investigations) | 6 | 0
Alanine aminotransferase increased (Investigations) | 10 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 20 | 0
Creatinine increased (Investigations) | 6 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 26 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 0
Hypokalemia (Metabolism and nutrition disorders) | 11 | 3
Hyponatremia (Metabolism and nutrition disorders) | 13 | 0
Metabolic/Laboratory-other (Investigations) | 7 | 0
Dizziness (Nervous system disorders) | 9 | 0
Depression (Psychiatric disorders) | 4 | 0
Neuropathy-sensory (Nervous system disorders) | 28 | 10
Vision-blurred (Eye disorders) | 5 | 0
Abdomen, pain (Gastrointestinal disorders) | 6 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 10 | 0
Head/headache (Nervous system disorders) | 7 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less